CLINICAL TRIAL: NCT06056479
Title: Efficacy Of Ultrasound Guided External Oblique Intercostal Plane Block for Postoperative Analgesia in Patients Undergoing Subcostal Nephrectomy: A Randomised Trial
Brief Title: Efficacy Of Ultrasound Guided External Oblique Intercostal Plane Block for Subcostal Nephrectomy
Acronym: EOINB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amal Gouda Elsayed Safan, lecturer of anaethesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9/2023ANET1-1
Record Dates: First submitted 2023-09-11; First posted 2023-09-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- external oblique intercostal block after induction (Active Comparator): After induction of general anesthesia, external oblique intercostal blocks will be performed with patients positioned in the supine position with their ipsilateral arm abducted.
  Initially the probe is placed in a cephalad to caudad paramedian direction at the anterior axillary line, and the external oblique muscle identified at the level ribs 6 and 7 in line with the xiphoid process. To confirm correct identification of the external oblique muscle, With 17gauge echogenic ultrasound needle will be advanced in plane from a superomedial-to-inferolateral direction, through the external oblique muscle.30 ml of bupivacaine 0.25% will be administered incrementally.
  Interventions: Procedure: external oblique intercostal block
- postoperative morphine per patient request (No Intervention): In this group no block will be done only morphine will be given intraoperatively- according to hemodynamic change and postoperative by morphine per patient request

INTERVENTIONS:
Procedure: external oblique intercostal block — 20 ml of bupivacaine 0.25% will be administered by US into external oblique intercostal plane at the level of sixth rib space .
  Arms: external oblique intercostal block after induction

SUMMARY:
The patients will be randomly allocated into two equal groups using a computer program.

Group A: will receive external oblique intercostal block after induction. Group B: will receive postoperative morphine per patient request.

DETAILED DESCRIPTION:
General anaesthesia induction will be achieved using fentanyl 1µg/kg (IV), propofol 2mg/kg (IV), and0.5mg/kg of IV Atracurium. General anaesthesia will be maintained with mechanical ventilation with isoflurane with O2 \ Air mixture.

During anaesthesia maintenance Intraoperatively, if BP or heart rate (HR) increase more than 20% from baseline, intravenous morphine will be given to stabilize the patients' haemodynamics.

All patients will receive 1g intravenous paracetamol and 4mg ondansetron 8mg dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

- Eligible patients will be older than 18 years old with American society of anestheologist ASA physical status I, II and III scheduled for Trans-Abdominal ( Anterior Subcostal) Nephrectomy

Exclusion Criteria:

* Patients who are:
* Unable to cooperate.
* Patients who have allergy to any of the study drugs.
* Patients who are on opioids.
* Known abuse of alcohol or medication.
* Local infection at the site of injection or systemic infection.
* Pregnancy
* Patients with coagulation disorders or on anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Time for first rescue analgesia | day 0
  hours

SECONDARY OUTCOMES:
VAS score | 24 hours
  1 to 10 (0 is interpreted as no pain, 1-4 mild pain, 5-6 moderate pain, 7-10 severe pain)
rescue analgesics | 24hous
  morphine mg

CONTACTS AND LOCATIONS:
Overall Officials: AMAL G SAFAN, MD, Principal Investigator — Menoufia University
Locations (1):
- Menoufia university, Cairo, Shibin Elkom, Egypt

IPD SHARING:
Plan to Share IPD: No